CLINICAL TRIAL: NCT06921876
Title: Autistic Eye Contact? A Hermeneutic Phenomenological Multicenter Study on Experiences With Eye Contact Between Adults With and Without Autism Spectrum Disorder With Use of Semi-structured Interviews. Using Semi-structured Interviews, the Experiences of People With and Without Autism Regarding Eye Contact Were Made Clear. The Topic List for These Semi-structured Interviews Was Developed in Co-design With People With Autism.
Brief Title: Autistic Eye Contact?
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Dimence Groep (Unknown)
Responsible Party: Principal Investigator, Jos Boer, MSc, UMC Utrecht
Other Study IDs: 55990; Dimence Groep (Other: Dimence Groep)
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder (ASD); Neurotypical
Keywords: Autism Spectrum Disorder; ASD; Neurotypical; Eye contact; Experience; Qualitative research
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Autism: The group of adults with ASD consisted of participants who were receiving outpatient treatment at one of three specialized centers for ASD, located in Deventer, Rotterdam or Amsterdam in the Netherlands.
- Neurotypicals: The group of adults without ASD consisted of participants who were never diagnosed with autism and lived in the Netherlands.

SUMMARY:
This research explored both breadth and depth of the experiences with eye contact in adults with and without ASD. A hermeneutic phenomenological multicenter design was used in which 15 adults with ASD and 15 adults without ASD were interviewed, using semi-structured interviews. Analyses using Multisite Qualitative Analysis (MSQA) and PRICE-model for saturation.

DETAILED DESCRIPTION:
This study aimed to examine the subjective eye contact experiences of adults with ASD compared to adults without ASD. Factors such as beliefs about the phenomenon, problems because of eye contact, development in eye contact, interpretations of others and more were explored.

To get insight in the subjective eye contact experiences of adults with ASD compared to adults without ASD, a hermeneutic phenomenological design using Multisite Qualitative Analysis (MSQA) and the PRICE-model for saturation during data analysis were used. MSQA enables the highest qualitative accuracy, the gathering of rich context-specific insights and maximizing the applicability. Semi-structured interviews was chosen for data collection and analysis because adults with ASD attach importance to on the one hand having the space to share their experiences in their own way, but on the other hand need frameworks to know what is asked of them. Hermeneutic phenomenological approach, grounded in philosophical concepts developed by Heidegger and Gadamer, made it possible to create meaning on how people experience a situation or phenomenon, such as eye contact, in a flexible and practical way.

Multisite design was chosen in response to criticism that single-site findings would limit the relevance and transferability and reliability to other settings. The Consolidated criteria for reporting qualitative studies (COREQ) checklist was used for reporting the research data. For the checklist. In addition, the Standards for Reporting Qualitative Research (SRQR) checklist was used. The research design was developed in collaboration with three adults with ASD and three adults without ASD, in order to include relevant information from the perspective of the target groups.

The semi-structured interviews were conducted using a topic list. This topic list consisted of the following sub questions:

Meaning:

* What do you think is the meaning of the term eye contact?
* In your opinion, are there different ways of making eye contact? If so, which?
* What do you think about the opinion that eye contact is abnormal in autism?

Development:

* Was the subject of eye contact brought up in your youth? If so, how?
* Did you learn how to make eye contact?
* Does your experiences with eye contact influenced how you lived your life? How?

Initiative to eye contact:

* Does it matter to you how others make eye contact with you? Why?
* Does the way you make eye contact with others depend on the situation or the person? Why?
* Do you adjust your eye contact to situations and/or people?

Interpretation of eye contact:

* Are there for you different ways of having eye contact? Which one?
* Are there for you different meanings of eye contact? Which one?

Dealing with eye contact:

* How do you make eye contact when interacting with others? Does that happen automatically?
* Do you consciously think about having eye contact? How come?
* How do you experience having eye contact with others? How come?

Wishes:

Would you like your eye contact with others to be different?/Do you need to improve the eye contact you have with others? If not, why? If so, why?

ELIGIBILITY:
Adults with autism

Inclusion criteria

* Diagnosed with autism according to an internationally recognized classification system
* Receiving outpatient treatment at a specialized autism center in the Netherlands
* Being able to understand the themes to be discussed
* Motivation to participate in the research

Exclusion criteria

* Insufficient command of the Dutch language
* Use of alcohol and/or recreational drugs during the study
* Too much mental instability to participate in the study
* Familiarity with treatment in intellectual disability care

Adults without autism

Inclusion criteria

* Being able to understand the themes to be discussed
* Motivation to participate in the research

Exclusion criteria

* Insufficient command of the Dutch language
* Use of alcohol and/or recreational drugs during the study
* Too much mental instability to participate in the study
* Familiarity with treatment in intellectual disability care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Experiences with eye contact with use of semi-structured interviews | June to September 2024
  The subjective eye contact experiences of adults with ASD compared to adults without ASD, using semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Nynke Boonstra, Professor, Study Chair — UMC Utrecht
Locations (1):
- Dimence Groep, Deventer, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No
On request.